CLINICAL TRIAL: NCT05601310
Title: 12,13-DHOME and Noradrenaline Are Associated With Occurrence of Acute Myocardial Infarction in Patients With Type 2 Diabetes Mellitus: A Untargeted Metabolomics Study
Brief Title: Metabolic Characteristics of Type 2 Diabetes Mellitus Combined With Acute Myocardial Infarction: A Untargeted Metabolomics Study
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Weiping Li, chief physician, Beijing Friendship Hospital
Other Study IDs: BFH-Metabolomics and STEMI
Record Dates: First submitted 2022-10-18; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: STEMI
Keywords: STEMI; Metabolomics; Biomarkers; Type 2 Diabetes Mellitus
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Diabetes Mellitus, Type 2 | interventions — Liquid Chromatography-Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: in the group, the participants exhibited negative results or <50% obstruction upon coronary artery CT or coronary angiography. The group did not have coronary heart disease and diabetes
  Interventions: Device: liquid chromatography-mass spectrometry (LC/MS) analysis
- T2DM group: in the group, the participants exhibited negative results or <50% obstruction upon coronary artery CT or coronary angiography. The group did not have coronary heart disease but have type 2 diabetes mellitus.
  Interventions: Device: liquid chromatography-mass spectrometry (LC/MS) analysis
- T2DM+AMI group: In the group, we eventually recruited 30 adult patients who were firstly diagnosed ST-elevation myocardial infarction (STEMI) within 12 hours of appearance chest pains or other AMI symptoms and had no previous history of coronary artery disease (CAD). Peripheral venous blood samples were drawn from subjects on admission or prior to coronary revascularization.
  Interventions: Device: liquid chromatography-mass spectrometry (LC/MS) analysis

INTERVENTIONS:
Device: liquid chromatography-mass spectrometry (LC/MS) analysis — To obtain a complete metabolic profile, untargeted metabolomics analysis was conducted by using UPLC-MS. Chromatographic separation was accomplished in an Thermo Vanquish system equipped with an ACQUITY UPLC®HSS T3 (150×2.1 mm, 1.8 µm, Waters, USA) column maintained at 40 ℃. The temperature of the autosampler was 8 ℃. The ESI-MSn experiments were executed on the Thermo Q Exactive mass spectrometer with the spray voltage of 3.5 kV and -2.5 kV in positive and negative modes, respectively. The capillary temperature was 325℃. The analyzer scanned over a mass range of m/z 81-1 000 for full scan at a mass resolution of 70 000. The normalized collision energy was 30 eV(19606840). The detected ions were all under isotopic calibration with the accurate masses of the reference standards.

SUMMARY:
This study is a retrospective case-control study. In this study, through untargeted metabolomics, investigators identified several specific changed serum metabolites in T2DM patients with or without AMI and their functions/category. Moreover, researchers selected several endogenous candidate biomarkers with larger fold change for validation in expanded population to find biomarkers which effectively predict the development of STEMI in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients meet the diagnostic criteria of "Guidelines for the Diagnosis and Treatment of Acute ST-segment Elevation Myocardial Infarction (2015)".
* STMEI patients undergoing emergency PCI should undergo emergency PCI within 12 hours of onset at Beijing Friendship Hospital affiliated to Capital Medical University.
* All diabetic patients meet the diagnostic criteria for type 2 diabetes.
* They agreed to be enrolled in the trial and signed the informed consent.

Exclusion Criteria:

* Combined with severe valvular disease or congenital heart disease, hypertension, chronic kidney disease, stroke, hyperlipidemia, previous history of coronary artery disease.
* Involved in acute infection, severe hepatic dysfunction, tumor, rheumatic immune disease.
* Incomplete clinical information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ① Patients with acute ST-segment elevation myocardial infarction (STEMI) who underwent emergency PCI in Beijing Friendship Hospital (Xicheng District) affiliated to Capital Medical University. ②In the Beijing Friendship Hospital (Xicheng District) affiliated to Capital Medical University, coronary angiography showed negative coronary angiography or coronary artery CT showed <50% obstruction in patients with non-coronary heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
There are differences in the metabolic profile of diabetic patients with or without combined acute myocardial infarction | December 16th, 2020
  About 10ml of venous blood was collected on the admission, serum was separated. To obtain a complete metabolic profile, untargeted metabolomics analysis was conducted by using UPLC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Li, MD, Study Director — Beijing Friendship Hospital
Locations (1):
- Weiping Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No